CLINICAL TRIAL: NCT02238132
Title: Postmarketing Surveillance Study (as Per §67(6)AMG[German Drug Law]) of Atrovent® Inhalets in Chronic Obstructive Airways Disease
Brief Title: Postmarketing Surveillance Study of Atrovent® Inhalets in Chronic Obstructive Airways Disease
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 244.2491
Record Dates: First submitted 2014-09-11; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Chronic Obstructive Airways Disease
  Interventions: Drug: ATROVENT® inhalets

INTERVENTIONS:
Drug: ATROVENT® inhalets

SUMMARY:
To obtain further information on the tolerability of Atrovent® inhalets in the treatment of Chronic Obstructive Airways Disease under conditions of daily practice

ELIGIBILITY:
Inclusion Criteria:

* Primarily, Patients with chronic obstructive airways disease
* Only patients who had not been treated with Atrovent® in the last year were to be considered for inclusion

Exclusion Criteria:

- Contraindications listed in the Instructions for Use/Summary of Product Characteristics for Atrovent® inhalets

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic obstructive airways disease recruited at general practitioners, pneumologists, internists
Sampling Method: Non-Probability Sample
Enrollment: 374 (Actual)
Dates: Start 1998-12; Primary Completion 1999-11 (Actual)

PRIMARY OUTCOMES:
Investigator assessment of improvement in the clinical picture of the course on a 6-point symptoms profile | Up to 4 weeks after first study drug administration

SECONDARY OUTCOMES:
Investigator assessment of efficacy on a 4-point scale | Up to 4 weeks after first study drug administration
Investigator assessment of tolerability on a 4-point scale | Up to 4 weeks after first study drug administration
Number of patients with adverse drug reactions | Up to 4 weeks after first study drug administration
Number of patients who withdrew from the study | Up to 4 weeks after first study drug administration
Number of patients who changed the concomitant medication | Up to 4 weeks after first study drug administration
Number of patients who continued the treatment | Up to 4 weeks after first study drug administration
Patient assessment of efficacy on a 4-point scale | Up to 4 weeks after first study drug administration
Patient assessment of tolerability on a 4-point scale | Up to 4 weeks after first study drug administration